CLINICAL TRIAL: NCT01698905
Title: A Phase II, Single Arm, Open Label Study of Treatment-free Remission in Chronic Myeloid Leukemia (CML) Chronic Phase (CP) Patients After Achieving Sustained MR4.5 on Nilotinib
Brief Title: Treatment-free Remission After Achieving Sustained MR4.5 on Nilotinib (ENESTop)
Acronym: ENESTop
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2408; 2012-003186-18 (EudraCT Number)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: AMN107; CML; Phase II; single arm; open label; nilotinib; treatment-free remission; MR4.5; confirmed loss of MR4; loss of MMR; Ph+ CML-CP
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nilotinib (Experimental): Patients with minimum 3 years of tyrosine kinase inhibitor treatment (first with imatinib and then switched to nilotinib) since initial diagnosis, at least 2 years of nilotinib treatment prior to study entry and who achieved MR4.5 (local laboratory assessment) during nilotinib treatment, and determined by a Novartis designated central PCR lab assessment at screening
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — Nilotinib was dosed by weight or body surface area.
  Nilotinib 300 mg BID or 400 mg BID was be administered orally at approximately 12 hour intervals, and must not have been taken with food. The capsules were to be swallowed whole with water.
  No food should have been consumed for at least 2 hours before the dose was taken and no additional food should have been consumed for at least one hour after the dose was taken. Patients were also allowed to enter this study on the same dose they were taking prior to study entry. Patients who required permanent dose reduction from their original starting dose were to be allowed to enter this study on the same dose only if the patient maintained this dose for a minimum of 6 months prior to study entry.
  Other Names: AMN107

SUMMARY:
A clinical research study to find out if it is safe to stop the drug nilotinib (Tasigna) in chronic myeloid leukemia (CML) patients. Patients who started treatment with imatinib (Gleevec) when they were first diagnosed with CML, then switched to nilotinib (Tasigna) for at least 2 years with the combined time on imatinib (Gleevec) and nilotinib (Tasigna) for at least 3 years and have very small amount of leukemia cells remaining after the nilotinib (Tasigna) treatment will qualify for the study.

DETAILED DESCRIPTION:
The Primary objective was to evaluate the proportion of patients in TFR within 48 weeks following nilotinib cessation.

This study originally consisted of seven phases (five treatment phases and two treatment-free phases) from which two were the focus of this primary analysis report (consolidation, TFR and treatment re-initiation) The study consisted of 2 main phases: Consolidation and TFR

Nilotinib treatment consolidation phase (NTCS): Patients who satisfied all inclusion/exclusion criteria were enrolled in the consolidation phase and continued to receive nilotinib for 52 weeks at the dose which the patient was receiving prior to study entry. If a patient maintained MR4.5 throughout the consolidation phase, he/she was eligible to enter in the TFR phase. If a patient had confirmed loss of MR4.5 during the consolidation phase, he/she was not eligible to enter in the TFR phase and continued nilotinib treatment.

Nilotinib TFR phase: Patients who were eligible to enter in the TFR phase after completing the 52 week consolidation phase stopped taking nilotinib on the first day of the TFR phase. Duration of this phase was up to 520 weeks after the last patient enters in the TFR phase.

Nilotinib treatment re-initiation phase (NTRI): If a patient had a confirmed loss of MR4 (two consecutive BCR-ABL >0.01% IS) or loss of MMR (BCR-ABL >0.1% IS) in the TFR phase, the patient restarted nilotinib treatment. Patients will be on nilotinib treatment for up to 520 weeks after the last patient entered the nilotinib TFR phase, or until a patient experience unacceptable toxicity, disease progression and/or treatment discontinued at the discretion of the Investigator or if the patient withdrew consent. Nilotinib cessation was not attempted for a second time in the patient who reinitiated treatment or discontinued following the TFR phase.

Nilotinib treatment continuation phase (NTCT) and Nilotinib treatment prolonged continuation phase (NTCT-P): Patients who were not eligible to enter into the TFR phase after completing the 52-week NTCS phase entered the nilotinib treatment continuation (NTCT) phase and would continue treatment with nilotinib for another 52 weeks (a total of 104 weeks of treatment). Patients who were not able to maintain MR4.5 and had a confirmed loss of MR4.5 during the NTCT phase were not eligible to enter the TFR-2 phase. These patients entered into the nilotinib prolonged treatment continuation phase (NTCT-P) and continued nilotinib treatment until 520 weeks after the last patient entered the nilotinib TFR phase, or until the patients experience unacceptable toxicity, disease progression and/or treatment would be discontinued at the discretion of the Investigator or withdrawal of consent.

Nilotinib TFR-2 phase: Patients who maintained MR4.5 during the NTCT phase were eligible to cease nilotinib treatment and enter the TFR-2 phase. The duration of the nilotinib TFR-2 phase is up to 520 weeks after the last patient entered the TFR phase. Patients stopped taking nilotinib therapy on the day they entered the TFR-2 phase.

Nilotinib treatment re-initiation-2 (NTRI-2): If a patient had a loss of MMR or a confirmed loss of MR4 during the TFR-2 phase, he/she entered the nilotinib treatment re-initiation-2 (NTRI-2) phase and resumed nilotinib treatment at a dose of either 300 mg or 400 mg bid.

Safety follow-up was performed within 30 days after the last dose of study treatment or the last day in TFR/TFR-2.

Post-treatment follow-up visits were performed every 12 weeks up to 520 weeks after the last patient entered the nilotinib TFR phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients >= 18 years of age
2. ECOG Performance Status of 0, 1, or 2
3. Patient with diagnosis of BCR-ABL positive CML CP
4. Patient has received a minimum of 3 years of tyrosine kinase inhibitor treatment (first with imatinib (> 4 weeks) and then switched to nilotinib) since initial diagnosis
5. Patient has at least 2 years of nilotinib treatment prior to study entry.
6. Patient has achieved MR4.5 (local laboratory assessment) during nilotinib treatment, and determined by a Novartis designated central PCR lab assessment at screening
7. Adequate end organ function as defined by:

   * Direct bilirubin ≤ 1.5 x ULN except for i) patient with documented Gilbert's syndrome for whom any bilirubin value is allowed and ii) for patients with asymptomatic hyperbilirubinemia (liver transaminases and alkaline phosphatase within normal range)
   * SGOT(AST) and SGPT(ALT) < 3 x ULN (upper limit of normal)
   * Serum lipase ≤ 2 x ULN
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Serum creatinine < 1.5 x ULN
8. Patients must have the following electrolyte values ≥ LLN (lower limit of normal) limits or corrected to within normal limits with supplements prior to the first dose of study medication:

   * Potassium
   * Magnesium
   * Total calcium (corrected for serum albumin)
9. Patients must have normal marrow function as defined below:

   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
   * Platelets ≥ 100 x 109/L
   * Hemoglobin ≥ 9.0 g/dL
10. Written informed consent obtained prior to any screening procedures

Exclusion Criteria:

1. Prior AP, BC or allo-transplant
2. Patient has documented MR4.5 at the time when switched from imatinib to nilotinib
3. Patients with known atypical transcript
4. CML treatment resistant mutation(s) (T315I, E255K/V, Y253H, F359C/V) detected if a testing was done in the past (there is no requirement to perform mutation testing at study entry if it was not done in the past)
5. Dose reductions due to neutropenia or thrombocytopenia in the past 6 months
6. Patient ever attempted to permanently discontinue imatinib or nilotinib treatment
7. Known impaired cardiac function including any one of the following:

   * Inability to determine the QT interval on ECG
   * Complete left bundle branch block
   * Long QT syndrome or a known family history of long QT syndrome
   * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia
   * QTcF > 480 msec
   * History or clinical signs of myocardial infarction within 1 year prior to study entry
   * History of unstable angina within 1 year prior to study entry
   * Other clinically significant heart disease (e.g. uncontrolled congestive heart failure or uncontrolled hypertension)
8. Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes (defined as HbA1c > 9%), uncontrolled infection)
9. History of acute pancreatitis within 1 year prior to study entry or past medical history of chronic pancreatitis
10. Known presence of a significant congenital or acquired bleeding disorder unrelated to cancer
11. History of other active malignancy within 5 years prior to study entry with the exception of previous or concomitant basal cell skin cancer, previous cervical carcinoma in situ treated curatively
12. Patients who have not recovered from prior surgery
13. Treatment with other investigational agents (defined as not used in accordance with the approved indication) within 4 weeks of Day 1
14. Patients actively receiving therapy with strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to study entry. See Appendix 14.1 for a list of these medications. This list may not be comprehensive.
15. Patients actively receiving therapy with herbal medicines that are strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to study entry. These herbal medicines may include Echinacea, (including E. purpurea, E. angustifolia and E. pallida), Piperine, Artemisinin, St. John's Wort, and Ginkgo.
16. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either safely discontinued or switched to a different medication prior to study entry. (Please see www.azcert.org/medical-pros/drug-lists/printable-drug-list.cfm for a list of agents that prolong the QT interval.)
17. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery)
18. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
19. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must have a negative serum pregnancy test before initiation of study treatment and must also use highly effective methods of contraception while enrolled in the study. The use of highly effective contraception should continue for at least 14 days after the last dose of study treatment or until the last day of TFR/TFR-2, or for the duration of a monthly cycle of oral contraception, whichever is longer. Acceptable forms of highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception, women should be stable on the same pill for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks prior to enrolling. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential. If a study patient becomes pregnant or is suspected of being pregnant during the study or within 30 days as part of safety evaluations after the final dose of nilotinib, the Study Doctor needs to be informed immediately and any ongoing study treatment with nilotinib has to be stopped immediately.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2015-11-26 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (59):
- United States (5):
  - USC Kenneth Norris Comprehensive Cancer Center, Los Angeles, California
  - Indiana Blood and Marrow Institute, Beech Grove, Indiana
  - St Agnes Hospital, Baltimore, Maryland
  - University of Texas Medical Branch, Galveston, Texas
  - Compass Oncology, Vancouver, Washington
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia (2):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Box Hill, Victoria
- Novartis Investigative Site, Antwerp, Belgium
- Brazil (6):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Rio de Janiero, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
- Canada (4):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (5):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Ulm
- Greece (3):
  - Novartis Investigative Site, Athens, Attica
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Athens
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Narita, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Chiba
- Novartis Investigative Site, Monterrey, Nuevo León, Mexico
- Poland (3):
  - Novartis Investigative Site, Krakow, Lesser Poland Voivodeship
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Warsaw
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Seocho Gu, South Korea
- Spain (6):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mahon FX, Boquimpani C, Kim DW, Benyamini N, Clementino NCD, Shuvaev V, Ailawadhi S, Lipton JH, Turkina AG, De Paz R, Moiraghi B, Nicolini FE, Dengler J, Sacha T, Takahashi N, Fellague-Chebra R, Acharya S, Wong S, Jin Y, Hughes TP. Treatment-Free Remission After Second-Line Nilotinib Treatment in Patients With Chronic Myeloid Leukemia in Chronic Phase: Results From a Single-Group, Phase 2, Open-Label Study. Ann Intern Med. 2018 Apr 3;168(7):461-470. doi: 10.7326/M17-1094. Epub 2018 Feb 20. PMID 29459949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 163 patients were enrolled into this study. 126 of the 163 patients who completed 52 weeks of nilotinib treatment in the NTCS phase entered the TFR phase and were part of the Full analysis Set (FAS).
Pre-assignment Details: Approximately 117 patients were planned to be enrolled into this study.
Groups:
- NTCS Phase: Patients with minimum 3 years of tyrosine kinase inhibitor treatment (first with imatinib and then switched to nilotinib) since initial diagnosis, at least 2 years of nilotinib treatment prior to study entry and who achieved MR4.5 (local laboratory assessment) during nilotinib treatment, and determined by a Novartis designated central PCR lab assessment at screening
Period: Overall Study
Arm/Group | NTCS Phase
Started | 163
Still on Study Phase | 0
TFR Phase | 126
NTRI Phase | 51
NTCT Phase | 26
TFR-2 Phase | 2
NTRI-2 Phase | 1
NTCT-P Phase Phase | 6
Completed (Completed = Completed 52 weeks of NTCS phase) | 152
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Physician Decision | 2
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 1
Not completed — Subject/guardian decision | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety Set: The safety set included all patients who received at least one dose of study medication in the Consolidation Phase.
Arm/Group | NTCS Phase
Number analyzed (Participants) | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (13.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 77
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 127
  Black | 6
  Asian | 23
  Native American | 1
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients in Treatment Free Remission (TFR) Within 48 Weeks
Description: TFR is defined as no confirmed loss of MR4 (Molecular response 4.0 log reduction from baseline) or loss of MMR (major molecular response) and no re-starting of nilotinib therapy within 12 months following cessation of nilotinib. Confirmed loss of MR4 is two consecutive BCR-ABL > 0.01% IS. Loss of MMR does not require confirmation. Percentage of patients in TFR is calculated by dividing the number of patients with no documented confirmed loss of MR4, no documented loss of MMR and no re-starting of nilotinib therapy in the first 48 weeks after starting nilotinib TFR phase by the number of patients who entered nilotinib TFR phase, and multiplied by 100.
Time Frame: First 48 weeks following nilotinib cessation.
Population: Full Analysis Set (FAS): FAS included all patients who entered the TFR phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NTCS Phase
Number analyzed (Participants) | 126
Percentage of participants | 57.9 [48.8 to 66.7]

2. Secondary Outcome: Percentage of Patients in Treatment Free Remission (TFR) Within 96, 144, 192, 264 Weeks and Within 6,7,8,9 and 10 Years
Description: TFR is defined as no confirmed loss of MR4 (molecular response 4.0 log reduction from baseline) or loss of MMR (major molecular response) and no re-starting of nilotinib therapy within 12 months following cessation of nilotinib. Confirmed loss of MR4 is two consecutive BCR-ABL > 0.01% IS. Loss of MMR does not require confirmation. Percentage of patients in TFR is calculated by dividing the number of patients with no documented confirmed loss of MR4, no documented loss of MMR and no re-starting of nilotinib therapy in the first 96, 144, 192, 264 weeks and within 6,7,8,9 and 10 years after starting nilotinib TFR phase by the number of patients who entered nilotinib TFR phase, multiplied by 100.
Time Frame: 96, 144, 192, 264 weeks and within 6,7,8,9 and 10 years following nilotinib cessation
Reporting Status: Not Posted, anticipated posting 2026-01

3. Secondary Outcome: Progression Free Survival (PFS) to Accelerated Phase/Blast Crisis (AP/BC) or Death
Description: Kaplan-Meier (KM) estimation of PFS. PFS is measured from the date of start of nilotinib TFR phase (cessation of nilotinib) to the date of the earliest of the event: progression to AP/BC, or death from any cause. Patients not known to have recurred or died on or before the cut-off date for the KM analysis will have their PFS interval right-censored at the earlier of the date of their last assessment (cytogenetic, hematology or extramedullary) for patients who are still on study and at the date of last contact for patients are in follow-up.
Time Frame: nilotinib cessation up to approximately 580 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

4. Secondary Outcome: Treatment Free Survival (TFS)
Description: Kaplan-Meier (KM) estimation of TFS is measured from the date of the start of the nilotinib TFR phase to the date of the earliest of the following: loss of MMR, confirmed loss of MR4, re-start of nilotinib treatment, progression to AP/BC or death from any cause. Patients not known to have had any of the events or died on or before the cut-off date for the KM analysis will have their TFS interval right-censored at the earlier of the date of their last assessment (PCR, cytogenetic, hematology or extramedullary) for patients who are still on study and at the date of last contact for patients are in follow-up. A TFS sensitivity analysis will be conducted by considering discontinuation from TFR phase due to any reason as an event, in addition to the events as defined above
Time Frame: nilotinib cessation up to approximately 580 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

5. Secondary Outcome: Overall Survival (OS)
Description: Kaplan-Meier (KM) estimation of OS. OS is measured from the date of start of nilotinib TFR phase to the date of death from any cause. If a patient is not known to have died, survival will be censored at the date of last contact.
Time Frame: nilotinib cessation up to approximately 580 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

6. Secondary Outcome: Change in BCR-ABL (Oncoprotein Product of BCR-ABL Fusion Gene) Transcripts After Re-start of Nilotinib Therapy
Description: Descriptive statistics of BCR-ABL over time after re-start of nilotinib therapy. ABL= Abelson leukemia virus and BCR=Break point cluster region
Time Frame: re-start of nilotinib up to approximately 48 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

7. Secondary Outcome: Percentage of Patients With Stable MMR in Nilotinib Re-initiation Phase
Description: Percentage of patients who are in stable MMR (stable MMR=BCR-ABL ≤ 0.1% IS) at 48, 96, 144, 192, 240, 288, 336, 384, and 432 weeks after achievement of that response in the nilotinib re-initiation phase for 48, 96, 144, 192, 240, 288, 336, 384, and 432 weeks is calculated by dividing the number of patients achieving MMR any time during the nilotinib re-initiation phase and having the same response at 48, 96, 144, 192, 240, 288, 336, 384, and 432 weeks after the first achievement of MMR, irrespective of whether there is loss of MMR in between, by the number of patients who achieved MMR at any time during the nilotinib re-initiation phase, and multiplied by 100.
Time Frame: start of nilotinib in re-initiation phase up to approximately 432 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

8. Secondary Outcome: Percentage of Patients With Stable MR4 in Nilotinib Re-initiation Phase
Description: Percentage of patients who are in stable MR4 (stable MR4=BCR-ABL ≤ 0.01% IS) at 48, 96, 144, 192, 240, 288, 336, 384, and 432 weeks after achievement of that response in the nilotinib re-initiation phase for 48, 96, 144, 192, 240, 288, 336, 384, and 432 weeks is calculated by dividing the number of patients achieving MR4 any time during the nilotinib re-initiation phase and having the same response at 48, 96, 144, 192, 240, 288, 336, 384, and 432 weeks after the first achievement of MR4, irrespective of whether there is loss of MR4 in between, by the number of patients who achieved MR4 at any time during the nilotinib re-initiation phase, and multiplied by 100.
Time Frame: start of nilotinib in re-initiation phase up to approximately 432 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

9. Secondary Outcome: Percentage of Patients With Stable MR4.5 in Nilotinib Re-initiation Phase
Description: Percentage of patients who are in stable MR4.5 (stable MR4.5=BCR-ABL ≤ 0.0032% IS) at 48, 96, 144, 192, 240, 288, 336, 384, and 432 weeks after achievement of that response in the nilotinib re-initiation phase for 48, 96, 144, 192, 240, 288, 336, 384, and 432 weeks is calculated by dividing the number of patients achieving MR4.5 any time during the nilotinib re-initiation phase and having the same response at 48, 96, 144, 192, 240, 288, 336, 384, and 432 weeks after the first achievement of MR4.5, irrespective of whether there is loss of MR4.5 in between, by the number of patients who achieved MR4.5 at any time during the nilotinib re-initiation phase, multiplied by 100.
Time Frame: start of nilotinib in re-initiation phase up to approximately 432 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until 30 days after the last dose of study treatment or the last day in the TFR/TFR-2 phase for approx. 35 months.
Description: Any sign or symptom that occurs during the study treatment plus 30 days post treatment.
Groups:
- TFR Phase: treatment-free remission
- NTRI Phase: nilotinib treatment re-initiation
- NTCT Phase: nilotinib treatment continuation
- TFR-2 Phase: treatment-free remission 2
- NTRI-2 Phase: nilotinib treatment re-initiation 2
- NTCT-P Phase: nilotinib treatment prolonged continuation
- All Patients: All patients enrolled in the study
Arm/Group | NTCS Phase | TFR Phase | NTRI Phase | NTCT Phase | TFR-2 Phase | NTRI-2 Phase | NTCT-P Phase | All Patients
All-Cause Mortality (participants affected / at risk) | 1/163 | 0/126 | 0/51 | 0/26 | 0/2 | 0/1 | 0/6 | 1/163
Serious Adverse Events (participants affected / at risk) | 21/163 | 8/126 | 4/51 | 3/26 | 0/2 | 0/1 | 0/6 | 34/163
Other Adverse Events (participants affected / at risk) | 80/163 | 70/126 | 29/51 | 11/26 | 0/2 | 0/1 | 2/6 | 122/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NTCS Phase (N=163) | TFR Phase (N=126) | NTRI Phase (N=51) | NTCT Phase (N=26) | TFR-2 Phase (N=2) | NTRI-2 Phase (N=1) | NTCT-P Phase (N=6) | All Patients (N=163)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NECROSIS (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3
DIVERTICULITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMATOLOGY TEST ABNORMAL (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
URETERIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
METRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
PLEURAL FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
ARTERIAL HAEMORRHAGE (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NTCS Phase (N=163) | TFR Phase (N=126) | NTRI Phase (N=51) | NTCT Phase (N=26) | TFR-2 Phase (N=2) | NTRI-2 Phase (N=1) | NTCT-P Phase (N=6) | All Patients (N=163)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 | 2 | 2 | 0 | 0 | 0 | 0 | 10
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 9
CONSTIPATION (Gastrointestinal disorders) | 5 | 0 | 3 | 0 | 0 | 0 | 0 | 8
DIARRHOEA (Gastrointestinal disorders) | 4 | 5 | 1 | 1 | 0 | 0 | 0 | 11
NAUSEA (Gastrointestinal disorders) | 5 | 2 | 4 | 1 | 0 | 0 | 0 | 9
FATIGUE (General disorders) | 6 | 3 | 3 | 1 | 0 | 0 | 0 | 12
NASOPHARYNGITIS (Infections and infestations) | 10 | 5 | 3 | 1 | 0 | 0 | 0 | 14
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 2 | 3 | 1 | 0 | 0 | 0 | 11
WEIGHT INCREASED (Investigations) | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 11
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 4
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 | 30 | 6 | 2 | 0 | 0 | 0 | 43
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 7
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 10 | 2 | 0 | 0 | 0 | 0 | 15
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 17 | 2 | 0 | 0 | 0 | 0 | 23
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 | 9 | 2 | 0 | 0 | 0 | 0 | 21
HEADACHE (Nervous system disorders) | 8 | 5 | 1 | 2 | 0 | 0 | 0 | 16
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 6
RASH (Skin and subcutaneous tissue disorders) | 7 | 1 | 4 | 0 | 0 | 0 | 0 | 12
HYPERTENSION (Vascular disorders) | 14 | 7 | 7 | 1 | 0 | 0 | 0 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.